CLINICAL TRIAL: NCT00067171
Title: Telephone Enhancement Procedure (TELE) for Continuing Care
Brief Title: Telephone Enhancement Procedure for Continuing Care - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Robert Hubbard, Ph.D., Duke University
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized
Other Study IDs: NIDA-CTN-0011-1
Record Dates: First submitted 2003-08-12; First posted 2003-08-13 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Substance-Related Disorders
Keywords: behavioral intervention
MeSH Terms: conditions — Substance-Related Disorders | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Behavior Therapy

SUMMARY:
The purpose of this study is to test a feasibility study of a telephone enhancement procedure (TELE) to improve participation in continuing care activities.

ELIGIBILITY:
Inclusion Criteria:

* Residential substance abuse treatment patients who reside within the pre-specified catchment area who complete continuing care plans prior to discharge.
* Voluntary admit to residential treatment center; substance abuse or dependence; reside in targeted counties; and may be reached by telephone.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339
Dates: Start 2003-01; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Treatment compliance, drug and alcohol astinence

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hubbard, Ph.D., Principal Investigator — Duke University
Locations (4):
- United States (4):
  - James Gilmore Jr. Treatment Center, Kalamazoo, Michigan
  - Julian F. Keith, Black Mountain, North Carolina
  - Walter B. Jones, ADATC, Greenville, North Carolina
  - Morris Village Alcohol & Drug Treatment Center, Columbia, South Carolina

REFERENCES:
- See also: Data Elements — http://www.ctndatashare.org/protocol-ctndatashare/new-protocols/nida-ctn-0011